CLINICAL TRIAL: NCT00095160
Title: Phase I, Open Label Safety, Pharmacokinetic, and Pharmacodynamic Dose Escalation/De-escalation Study of 852A Administered Intravenously to Subjects With Refractory Solid Organ Tumors
Brief Title: Safety Study of an Immune Response Modifier in Patients With Refractory Solid Organ Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Jeffrey Miller, M.D., Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003LS039; 1493-852A
Record Dates: First submitted 2004-11-01; First posted 2004-11-02 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms
Keywords: Solid Organ Tumors
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: 852A

SUMMARY:
Study 1493-852A is a phase 1 study with the primary objective of determining safety and the highest tolerated dose of an experimental immune response modifier administered intravenously to patients with solid organ tumors not responsive to currently available treatments. The secondary objective of the study is to monitor the tumor response to this form of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have solid organ tumors refractory to currently available treatments.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Have a life expectancy of 4 months
* Have normal organ and bone marrow function

Exclusion Criteria:

* Have had biologic, hormonal, anti-neoplastic chemotherapy, or radiation therapy within 4 weeks prior to the 1st dose of the study drug or those who have not recovered from adverse events from agents administered more than 4 weeks earlier.
* Use of investigational agent in the 4 weeks prior to 1st dose of the study drug
* Use of immunosuppressive therapy in the 4 weeks prior to the 1st dose
* Have a history of, or clinical evidence of, myocardial ischemia, congestive heart failure, or myocardial arrhythmias requiring treatment within the past 6 months
* Have uncontrolled intercurrent or chronic illness, but not limited to, ongoing or active infection such as hepatitis B or C, immune dysfunction such as autoimmune disease, endocrine dysfunction such as hypo- or hyperthyroidism, psychiatric illness such as depression or suicidal tendency or social situations that would limit compliance with study requirements
* Have a history of disease requiring ongoing steroid treatment
* Have a history of seizure disorders uncontrolled on medication
* Have a history of clinically significant coagulation or bleeding disorders or abnormalities
* Are HIV positive. HIV positive subjects are excluded from the study because of possible interactions with the immunomodulatory effects of 852A and because of potential pharmacokinetic interactions associated with combination retroviral therapy.
* Are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2003-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Safety and Pharmacokinetics

SECONDARY OUTCOMES:
Tumor Response

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States